CLINICAL TRIAL: NCT07151027
Title: Effectiveness Of Alcohol Addition In Ultrasound-Guided Periarticular Sacroiliac Joint Injection: A Double Blinded Randomized Prospective Study
Brief Title: Effectiveness Of Alcohol Addition In Ultrasound-Guided Periarticular Sacroiliac Joint Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Maged Shawky Farhat Gergis, Doctor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M797
Record Dates: First submitted 2025-08-18; First posted 2025-09-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sacro Iliac Joint Pain; Low Back Pain; Alcohol Induced Neurolysis
Keywords: Sacroiliatis; sacroiliac joint injection; prolotherapy; ethanol in low back pain; pain management
MeSH Terms: conditions — Low Back Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (group A) (Experimental): receives a mixture of alcohol 30%, dexamethasone and lidocaine 2%
  Interventions: Procedure: sacroiliac joint injection
- Active comparator group (group D) (Active Comparator): receives a mixture of dexamethasone and lidocaine 2%
  Interventions: Procedure: sacroiliac joint injection

INTERVENTIONS:
Procedure: sacroiliac joint injection — US-guided periarticular sacroiliac joint injection of a mixture of dexamethasone and lidocaine 2%
  Arms: Active comparator group (group D)
Procedure: sacroiliac joint injection — US-guided periarticular sacroiliac joint injection of a mixture of alcohol 30%, dexamethasone and lidocaine 2%
  Arms: Experimental group (group A)

SUMMARY:
The aim of this work is to evaluate the efficacy of adding alcohol to local anesthetics and steroids to provide pain relief in patients with sacroiliac joint pain.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common health problems globally. According to the Global Burden of Disease (GBD) Study 2021, low back pain is the leading cause of years lived with disability worldwide. It affects approximately 619 million people globally, and this number is projected to increase to 843 million by 2050 due to population growth and aging. (1) LBP may arise from multiple anatomical structures, such as muscle, intervertebral disc, fascia, and facet joint. Another common cause of LBP includes the sacroiliac joint (SIJ). It is estimated that around 10-38% of LBP cases originated from the SIJ. (2) In addition to its prevalence, SIJ pain lacks valid clinical/diagnostic tests and no therapeutic modalities for long-term improvement have been found yet. (3) Treatment of SIJ pain is another dilemma, and a wide range of therapeutic modalities has been used, including pharmacotherapy, chiropractic manipulation, SIJ injection (local anesthetics, steroid, or mixture), and surgical fixation. (4) Steroid and local anesthetic (LA) injections are widely used for managing SIJ pain, and evidence supports their effectiveness, particularly in the short to intermediate term but long-term benefit usually requires repeat injections or alternative treatments as radiofrequency or prolotherapy (5,6,7) Recently, alcohol neurolysis has gained popularity and become a well-established interventional technique in pain management, particularly for patients with chronic or cancer-related pain that is refractory to conventional therapies. (8)

Alcohol (Ethanol) in different concentrations (from 70% to 20%) has been used in different joints and pain syndromes such as trigeminal neuralgia, post-mastectomy pain syndrome, ankle pain from Morton neuroma and bursitis, and it proved its efficacy and safety. (9,10,11,12) Previous studies tried phenol injection in SIJ pain which acts nearly with the same mechanism of action as ethanol exerting a neurolytic effect through protein denaturation and nerve fiber destruction. Also proved its efficacy and safety. (13, 14) No previous studies used alcohol injection in SIJ.This study hypothesize that the use of alcohol (ethanol) 30% as an adjuvant to steroids and local anesthetics in SIJ as a novel approach may offer both short and long-term pain relief and reduce the frequency of repeated injections.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of either gender diagnosed with sacroiliac joint pain.
2. Patient aged 18-60 years old.
3. Patients with American Society of Anesthesiologists (ASA) physical status I-II.
4. Chronic pain at sacroiliac joint for more than 12 weeks.

Exclusion Criteria:

1. Patients with MRI confirmed other cause of Low back pain as (disc prolapse, spinal canal stenosis, etc.).
2. Patients without any positive provocative tests (FABER, Gaenslen's and Fortin's finger tests).
3. Patients had findings suggestive of another source of axial back pain.
4. Patients with symptoms radiating past the knee.
5. Patients with less than 5/5 strength in the lower extremity.
6. Patients with diminished reflexes.
7. Patients diagnosed with myelopathy, and positive neural tension signs including straight leg raise and/or slump test.
8. Obese patients (BMI ≥ 35 kg/m²).
9. Infection at the injection site.
10. Patients who have undergone previous spine or pelvic surgery.
11. Coagulation disorders as bleeding tendency and platelet dysfunction.
12. Allergy to local anesthetics.
13. Patients with mental disorders, as well as drug abuse.
14. Lumbar facet steroid injections within the past 12 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
Pain relief as measured by the visual analogue scale VAS scale | preoperative(baseline), immediate after injection, 4 weeks, 8 weeks, 4 months and 6 months after injection
  Presented by a 10 cm horizontal line representing the patient's pain intensity. Zero represents "no pain" while the upper limit (10 cm) represents the "worst pain imaginable.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | preoperative(baseline), immediate after injection, 4 weeks, 8 weeks, 4 months and 6 months after injection
  is a questionnaire designed to assess the degree of disability in low back pain. It comprises 10 sections, pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual activity, social life, and traveling. Each section is scored on a scale from 0 to 5, the total score is calculated by summing section scores, dividing by the maximum possible score, and multiplying by 100 to yield a percentage from 0 to 100% .with higher percentages denoting more severe disability. The total score is the number of questions with a positive response (yes) and reduction in four or more scores indicates that the treatment has achieved its goal.
Patient Satisfaction Score (PSS) | within 15 minutes after the procedure completion
  a self reported measure of a patient's overall satisfaction with care, a 5 point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied).
Time to first postoperative analgesic dose | interval (in hours) for the first 48 hours
  interval (in hours) from completion of the sacroiliac joint injection to the patient's first request for analgesia recorded by nursing staff then patient and his relatives after discharge. A longer time to first dose indicates more prolonged analgesic effect of the injection.
Cumulative Gabapentin consumption | 1 week, 4 weeks, 8 weeks, 4 months and 6 months after injection.
Procedure discomfort | within 15 minutes after the procedure completion
  Procedure discomfort via VAS scale
Complications | six months after injection
  I. Postoperative Nausea and Vomiting (PONV). II. Hyperalgesia III. Loss of Sensation IV. Lower Limb Muscle Weakness V. Infection at Injection Site

CONTACTS AND LOCATIONS:
Locations (1):
- FayoumU, Al Fayyum, Faiyum Governorate, Egypt